CLINICAL TRIAL: NCT06628258
Title: An Exploratory, Prospective, Open-Label, Interventional, Safety In-Use, Tolerability and Efficacy Study of Test Product "Moiz Cleansing Lotion" in Healthy Human Subjects.
Brief Title: A Clinical Study to Assess the Safety and Effectiveness of Test Product "Moiz Cleansing Lotion" in Healthy Adult Human Subjects With Varied Skin Types. (Dry, Oily, Sensitive, Mixed, Normal)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Collaborators: Glowderma Lab Private Limited (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NB240043-GL
Record Dates: First submitted 2024-09-14; First posted 2024-10-04 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: All Skin Types

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dry, sensitive, oily, mixed, normal skin type (Experimental): Test Product Name: Moiz Cleansing Lotion Product By: Glowderma Lab Private Limited Mode of Usage: Apply 5-10 ml of Moiz Cleansing Lotion to wet skin. Massage gently for 1-2 minutes, then rinse and pat dry.
  Frequency: Twice a Day Route of Administration: Topical.
  Interventions: Other: Moiz Cleansing Lotion

INTERVENTIONS:
Other: Moiz Cleansing Lotion — Mode of Usage: Apply 5-10 ml of Moiz Cleansing Lotion to wet skin. Massage gently for 1-2 minutes, then rinse and pat dry.
  Frequency: Twice a Day Route of Administration: Topical.

SUMMARY:
This is an exploratory, prospective, open-label, interventional, safety in-use, tolerability and efficacy study of the test product "Moiz Cleansing Lotion" in healthy human subjects.

DETAILED DESCRIPTION:
27 subjects with different skin type (dry/ oily/ sensitive/ mixed/) of either gender aged between 18 to 65 years old (both inclusive) at time consent will be enrolled to complete 25 subjects/test product in the study.

The potential subjects will be screened as per the inclusion & exclusion criteria only after obtaining written informed consent from the subjects. Subjects will be pre-screened by the screening department of NovoBliss Research. Subjects will be called telephonically by the recruiting department prior to the enrolment visit. Subjects will be told during screening (prior to enrolment) not to wear any facial make-up on the study visit day. The adult female subjects will be instructed to visit the facility as per the below visits-

* Visit 01 (Day 01): Screening, Enrolment, Baseline Evaluation, On Site Product Usage, Post Usage Evaluation.
* Visit 02 (Day 15 +2 Days): Product Usage Period, Evaluations
* Visit 03 (Day 30 +2 Days): Evaluations, End of Study

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 65 years (both inclusive) at the time of consent.
* Sex: Healthy male and non-pregnant/non-lactating females (Preferably equal).
* Females of childbearing potential must have a self-reported negative pregnancy test.
* Subject are generally in good health.
* Subject with dry, oily, mixed, sensitive and normal skin at a time of screening. (Dermatological Assessment)
* Subjects forearm must be free of cuts, tattoos, scratches, abrasions, scars, uneven skin tone, sunburn, excessive tan, excessive hair or open wounds on or near the test sites
* Subject is able to remain on stable doses of contraceptive or replacement hormonal therapy, including no therapy, 6 weeks prior to and for the duration of the study.
* If the subject is of childbearing potential, is practicing and agrees to maintain an established method of birth control (IUD, hormonal implant device/injection, regular use of birth control pills or patch, diaphragm, condoms with spermicide or sponge with spermicidal jelly, cream or foam, partner vasectomy or abstinence). Females will be considered as non-childbearing potential if they are surgically sterile, have been post-menopausal for at least 1 year or have had a tubal ligation.
* Subjects are willing to give written informed consent and are willing to come for regular follow up.
* Subjects who commit not to use medicated skincare products other than the test product for the entire duration of the study.
* Subject who have not participated in a similar investigation in the past three months.
* Willing to use test product throughout the study period.

Exclusion Criteria:

* History of any dermatological condition of the skin diseases.
* Subject with present condition of allergic response to any cosmetic product.
* Subject having allergic response to the ink.
* Subjects under chronic medication (e.g. aspirin-based products, anti-inflammatories, anti-histamines, corticotherapy etc.) that might influence the outcome of the study.
* Subject having acne of severe incidence (presence of nodules, cysts or numerous pustules) which requires pharmaceutical or cosmeceuticals, herbal product.
* Subjects who have applied topical product for at least 4 weeks and any systemic product for at least 3 months, before they participated in the study.
* History of alcohol or drug addiction.
* Subjects using other marketed products during the study period.
* Any other condition which could warrant exclusion from the study, as per the dermatologist's/investigator's discretion.
* Pregnant or breastfeeding or planning to become pregnant during the study period.
* History of chronic illness which may influence the cutaneous state.
* Subjects participating in other similar cosmetics, devices or therapeutic trials or skincare products within the last four weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2024-10-23 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
change in L*, a*, b* value by using Skin Colorimeter | before usage of the test product on Day 01 and after usage of the test product at T20 minutes on Day 01, Day 15 and Day 30.
  To evaluate the effectiveness of the test product in terms of change in L*, a*, b*
change in skin impurities using Visiopor® PP34N | before usage of the test product on Day 01 and after usage of the test product at T20 minutes on Day 01, Day 15 and Day 30.
  To evaluate the effectiveness of the test product in terms of change in skin impurities

SECONDARY OUTCOMES:
change in skin hydration using Corneometer CM 825 | before usage of the test product on Day 01 and after usage of the test product at T20 minutes on Day 01, Day 15 and Day 30.
  To evaluate the effectiveness of the test product in terms of change in skin hydration
change in skin barrier function using TEWAMeter | before usage of the test product on Day 01 and after usage of the test product at T20 minutes on Day 01, Day 15 and Day 30.
  To evaluate the effectiveness of the test product in terms of change in skin barrier function
change in overall dry skin score by dermatological evaluations | before usage of the test product on Day 01 and after usage of the test product at T20 minutes on Day 01, Day 15 and Day 30.
  To evaluate the effectiveness of the test product in terms of change in overall dry skin score where, 0: means absent and 4 means: Dominated by large scales, advanced roughness, redness present, eczematous changes and cracks
change in PGA score by dermatological evaluations | before usage of the test product on Day 01 and after usage of the test product at T20 minutes on Day 01, Day 15 and Day 30.
  To evaluate the effectiveness of the test product in terms of change in PGA score where 0 means: No appearance and 8 means: Severe
change in product perception questionnaire | before usage of the test product on Day 01 and after usage of the test product at T20 minutes on Day 01, Day 15 and Day 30.
  6. To evaluate the effectiveness of the test product in terms of change in product perception questionnaire where 0 means: Dislike extremely and 9 means liked extremly
change in visual and tactile assessment of scaliness | before usage of test product on Day 01 and after usage of test product at T20 minutes on Day 01, Day 15 and Day 30.
  To evaluate the effectiveness of the test product in terms of change in scaliness where 0 means: Absent and 4 means: Extreme
change in visual and tactile assessment of roughness | before usage of test product on Day 01 and after usage of test product at T20 minutes on Day 01, Day 15 and Day 30.
  To evaluate the effectiveness of the test product in terms of change in roughness where 0 means: Absent and 4 means: Extreme
change in visual and tactile assessment of redness | before usage of test product on Day 01 and after usage of test product at T20 minutes on Day 01, Day 15 and Day 30.
  To evaluate the effectiveness of the test product in terms of change in redness where 0 means: Absent and 4 means: Extreme
change in visual and tactile assessment of itchiness | before usage of test product on Day 01 and after usage of test product at T20 minutes on Day 01, Day 15 and Day 30.
  To evaluate the effectiveness of the test product in terms of change in itchiness where 0 means: None and 4 means: Severe
change in visual and tactile assessment of dryness | before usage of test product on Day 01 and after usage of test product at T20 minutes on Day 01, Day 15 and Day 30.
  To evaluate the effectiveness of the test product in terms of change in dryness where 0 means: No Skin Dryness and 4 means: Extreme Xerosis
change in visual and tactile assessment of smoothness | before usage of test product on Day 01 and after usage of test product at T20 minutes on Day 01, Day 15 and Day 30.
  To evaluate the effectiveness of the test product in terms of change in smoothness where 0 means: Very rough and 4 means: Very smooth
change in skin irritation | before usage of test product on Day 01 and after usage of test product at T20 minutes on Day 01, Day 15 and Day 30.
  Safety of test product will be evaluated in terms of change in skin irritation by dermatological assessment
change in dryness | before usage of test product on Day 01 and after usage of test product at T20 minutes on Day 01, Day 15 and Day 30.
  Safety of test product will be evaluated in terms of change in dryness by dermatological assessment
change in breakouts | before usage of test product on Day 01 and after usage of test product at T20 minutes on Day 01, Day 15 and Day 30.
  Safety of test product will be evaluated in terms of change in breakouts by dermatological assessment
change in allergic reactions | before usage of test product on Day 01 and after usage of test product at T20 minutes on Day 01, Day 15 and Day 30.
  Safety of test product will be evaluated in terms of change in allergical reactions by dermatological assessment

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Nayan K Patel, Principal Investigator — NovoBliss Research Pvt Ltd
Locations (1):
- NovoBliss Research Pvt.Ltd, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No